CLINICAL TRIAL: NCT02393014
Title: Activité Physique et prévention de la Chute du Patient âGé hospItalisé en Court séjouR: Etude de faisabilité (AGIR)
Brief Title: Physical Activity and Fall Prevention in Geriatric Inpatients in Acute caRe: Feasibility Study
Acronym: AGIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-30
Record Dates: First submitted 2015-02-05; First posted 2015-03-19 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2015-02

CONDITIONS: Elderly
Keywords: 65 years old or older; hospitalized in; geriatrics

ARMS (3):
- Low fall risk (Experimental): low fall risk patients
  Interventions: Procedure: Simple physical exercises
- Medium fall risk (Experimental): medium fall risk patients
  Interventions: Procedure: Simple physical exercises
- High fall risk (Experimental): high fall risk patients
  Interventions: Procedure: Simple physical exercises

INTERVENTIONS:
Procedure: Simple physical exercises — 1. The participant must stay out of the bed 3 hours. This pre-required level prevents the occurrence of acute postural mismatch which can occur when elderly patients are bedridden and too long increases the risk of falling.
  2. The participant stands standing in static equilibrium to a chair holding the back of it for 2 minutes. Depending on the patient's abilities, the exercise will be done on both feet or one foot.
  3. The participant performs a transfer activity of sitting to standing repeated 5 times (FTSS test). According to the patient's abilities, the exercise will be done with physical assistance or not.

SUMMARY:
This study aims to evaluate the feasibility and the impact on physical performance and falls occurence among geriatric inpatients hospitalized in acute care unit.

DETAILED DESCRIPTION:
Having developed many tools to determine fall risk of 65 years and older patients, Angers University Hospital plans to develop a corrective action to prevent the occurrence of falls in this population.

This study aims to assess the feasibility of a physical activity program with 3 difficulty levels (depending on the patient's risk of falling): easy (low fall risk), moderate (average fall risk) and difficult (high fall risk).

The implementation process should be simply and fastly applicable in practice for routine care by paramedics.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years old and older
* Being hospitalized in geriatric acute care unit of Angers University Hospital.
* No contraindications to physical activity practice.
* No contraindications to standing station and sitting station.
* Participants having given and signed an informed participation consent. If the participant is unable to answer, we will retain the disagreement expressed by a trusted person.
* Being affiliated to French social security

Exclusion Criteria:

* Refusal of participation
* Persons aged under 65.
* Topics including hospitalization at the entrance should not exceed 3 days.
* Participation in concomitant clinical trial.
* Civil Protection Measures such as trusteeship, guardianship or backup justice underway.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 278 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants in each category of fall risk having realized 75% and more of the exercises of at least one of the three difficulty levels of the physical activity program | up to 15 months
  The feasibility of the interventions of each fall risk category is defined as "at least 80% of the participants of a category having completed 75% and more of the exercises".

SECONDARY OUTCOMES:
Change of number of patients having realized the Five Time Sit and Stand (FTSS) test. | up to 15 months
For the patients having achieved FTSS test, the realization time (in seconds). | up to 60 seconds
Measure (by the medical team) of the difficulty to set up and carry out the exercises | up to 20 days
  This measure will be assessed with a scale : "very easy" ; "easy" ; "feasible" ; "difficult" ; "impossible"
Time needed by the paramedical team to achieve the exercises | up to 20 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Angers, Maine et Loire, France

REFERENCES:
- [Derived] Noublanche F, Simon R, Ben-Sadoun G, Annweiler C. Physical Activity and Fall Prevention in Geriatric Inpatients in an Acute Care Unit (AGIR Study): Protocol for a Usability Study. JMIR Res Protoc. 2022 Jul 11;11(7):e32288. doi: 10.2196/32288. PMID 35816381